CLINICAL TRIAL: NCT04379258
Title: Epidemiological Analysis of the Mortality of Critically Ill Patients With the COVID-19 Admitted to the Intensive Care Unit: An Observational, Prospective and Multicenter Study
Brief Title: Analysis of Mortality of Critically Ill Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Collaborators: Hospital Universitario del Tajo (Unknown); Puerta de Hierro University Hospital (Other); Hospital de Henares (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario de Móstoles (Other); Hospital Universitario Severo Ochoa (Unknown); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Universitario Madrid Sanchinarro (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Universitario Infanta Cristina (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario de Torrejón (Unknown); Hospital Universitario La Paz (Other); Hospital Universitario 12 de Octubre (Other); Hospital Christus Muguerza Betania, Puebla, Mexico (Unknown); Hospital General de Mexico (Other Government); Hospital Regional 1º de Octubre ISSSTE Mexico (Unknown); Hospital Juarez de Mexico (Other Government); Hospital Gea Gonzalez Mexico (Unknown); Hospital Civil de Guadalajara (Other); Hospital Regional de alta Especialidad Ixta, Mexico (Unknown); Hospital Ángeles Tampico, Mexico (Unknown); Hospital de la Beneficiencia Espaañola, Tampico, Mexico (Unknown); Hospital Ángeles Tijuana, Mexico (Unknown); Hospital Universitario UANL, Mexico (Unknown); Hospital H+ Querétaro, Mexico (Unknown); Hospital General de Zona 1A Venados, Mexico (Unknown); Centro Médico ABC Observatorio, Mexico (Unknown); Hospital Christus Muguerza Alta Especialidad, Nuevo León, Mexico (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVID-UCI_Spain
Record Dates: First submitted 2020-04-22; First posted 2020-05-07 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-02

CONDITIONS: COVID-19; Critical Illness; Effectiveness; Outcome, Fatal
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The recent pandemic of the COVID-19 disease has caused a national health emergency due to its severity and the clinical and social consequences of the disease. Crude mortality in Spain is 9.2%. However, the causes of death of critically ill patients with COVID-19 are unknown. To date, no treatment has been shown to be effective for the 2019-SARS-CoV-2 infection is recommended. Supportive care and isolation are recommended for infected individuals. Currently, observational studies on critically ill patients with COVID-19 have small samples. The objective is to evaluate the incidence of mortality and morbidity in COVID-19 disease in this group of critically ill patients, as well as the risk factors associated with mortality and the effectiveness of the treatments used compassionately.

DETAILED DESCRIPTION:
Introduction The World Health Organization (WHO) has recently declared SARS-CoV-2 (COVID-19) disease as an international alarm public health emergency. This ongoing pandemic of COVID-19 disease is devastating, despite widespread implementation of control measures, which is creating a challenge for national healthcare. Since the beginning of the epidemic until the date of this project, more than 800,000 cases have been detected in the world, of which almost 214,000 have been detected in Spain.

The results of the recent analysis of clinical characteristics in a selected cohort of 1,099 COVID-19 patients throughout China have shown that up to 15% (173 / 1,099) developed severe disease according to the American Thoracic clinical criteria for severe community pneumonia. Society, and of these seriously ill patients, 20.6% presented as admission to Intensive Care Units (ICU) (33/173, 19%), or the use of mechanical ventilation, both invasive and non-invasive. invasive (81/173, 46%) or death (14/173, 8%).

In a retrospective study that included 52 critically ill patients with COVID-19 admitted to the Intensive Care Unit (ICU) from the Wuhan Jin Yin-tan Hospital (Wuhan, China), a 28-day mortality rate of 61% was found, although the causes of death of the patients included were not reported.

Nowaday, the crude mortality in Europe is 5.4% of reported cases, although it is important to be noted that this calculation is subject to multiple notification biases and due to the different diagnostic test policies in the countries, and probable differences in healthcare and demographic models between countries. Similarly, in Spain, mortality with 213,024 cases notified to the National Surveillance Network is 10.4%. Using modeling, a mortality has been estimated among hospitalized cases that could reach 14% (95% confidence interval [CI] 3.9% -32%). However, the mortality and causes of death of critically ill patients with COVID-19 in Spain are still unknown.

To date, no specific antiviral treatment that has been shown to be effective for the 2019-SARS-CoV-2 infection is recommended. Symptomatic and supportive care, along with respiratory and contact isolation, are recommended for infected individuals.

Selective digestive decontamination (SDD) is a prophylactic treatment for critically ill patients, mainly requiring invasive mechanical ventilation, based on an oropharyngeal paste and an enteral suspension containing antimicrobials (usually tobramycin, colistin, and an antifungal) and an intravenous antibiotic (usually a cephalosporin. second generation), administered during the first 4 days of ICU treatment. The goal of SDD is to prevent or eradicate, if present, the abnormal, oropharyngeal and intestinal transport of potentially pathogenic microorganisms, such as aerobic gram-negative bacilli (AGNB), methicillin-sensitive Staphylococcus aureus, in patients at risk of nosocomial infections. In critically ill patients, it has been demonstrated with a high level of evidence, that SDD prevents serious infections and reduces mortality. In an observational study in two hospitals in China, 51% of the patients developed a hospital-acquired infection and this incidence was associated with an increase in mortality. Therefore, the preventive strategy of SDD could be postulated as an alternative to reduce mortality and the incidence of infections in critically ill patients with COVID-19. However, this hypothesis has not been evaluated at the moment.

At the present time, observational studies focused on the clinical characteristics of critically ill patients with COVID-19 and the factors associated with their mortality have small sample sizes, making knowledge of the epidemiology of critically ill patients clearly insufficient. And what is more relevant, this scenario of lack of knowledge, when extrapolated to the situation of the current outbreak in Spain, places us in the need to describe the epidemiological manifestations of the COVI-19 in Spain in order to handle with safety and efficiency the challenge of the control and treatment of the outbreak in Spain of the COVID-19.

Specifically, the study will focus on critically ill patients with COVID-19 for two reasons:

They represent the cohort of patients with the highest use of material and professional resources in the health system.

Given the current moment of pandemic and healthcare challenge, it is therefore pertinent to conduct an epidemiological surveillance of COVID-19 disease to reliably define the incidence of mortality and morbidity in this group of patients, as well as the risk factors for infection by SARS-CoV-2 associated with mortality.

Objective The main objective is to evaluate the mortality of critically ill patients with COVID-19 admitted to the ICU, as well as to analyze the factors associated with mortality.

The secondary objectives:

To analyze the epidemiological characteristics of critically ill patients with confirmed COVID-19 in Spain.

To describe the usual clinical practice in the ICU of critically ill adult patients with COVID-19, to identify risk patterns and possible effectiveness or adverse effects of the treatments received.

To compare the mortality of critically ill patients with COVID-19 treated with SDD compared with those who do not received SDD.

To describe the cause of death of critically ill patients with COVID-19 received invasive mechanical ventilation.

Method Design: An observational, prospective and multicenter study will be carry out, envolving of 12 ICUs in Madrid (University Hospital of Getafe, as coordinating center; University Hospital Puerta de Hierro, University Hospital del Henares of Coslada, University Hospital of Torrejón, Hospital Universitario Ramón y Cajal, Hospital Infanta Cristina, Hospital del Tajo, Hospital Quirón Madrid Sanchinarro, Hospital Universitario Severo Ochoa, Hospital Universitario Gregorio Marañón, Hospital Universitario de Móstoles, Hospital Universitario La Princesa, Hospital Universitario La Paz, Hospital Universitario Doce de Octubre, and Hospital Santa Creu i Sant Pau in Barcelona). Inclusion criteria: patients over 18 years of age who are admitted to the ICU with the confirmed diagnosis of COVID-19.

Recruitment period: The study will start once the study has been approved by the Ethics and Research Committee of the Hospital Universitario de Getafe with an expected date of April 2020, with an estimated duration of 3 months.

Case definition: Any critically ill patients with a positive respiratory tract sample result (tracheal aspirate or nasopharyngeal exudate) using the PCR technique for the SARS-CoV-2 virus and requiring admission to the ICU at trial will be considered a confirmed case of COVID-19 of the physician in charge of the patient.

Data collection: Demographic variables: age, sex, reason for admission to the ICU.

Comorbidities: severity at ICU admission (SAPSIII); Daily SOFA until day 7, diabetes mellitus, high blood pressure, chronic obstructive pulmonary disease, other chronic lung diseases (interstitial lung disease), chronic kidney failure, previous liver disease (cirrhosis), immunosuppression, previous heart disease (ischemic, valvular), chronic arrhythmias (atrial fibrillation); previous cerebrovascular disease (ischemic or hemorrhagic).

Noninvasive respiratory support prior to ICU admission: non-invasive ventilation, or high flow therapy with nasal cannula, and duration of non-invasive respiratory support.

Invasive respiratory support parameters during the first 7 days: tidal volume, level of positive end-expiratory pressure, plateau pressure, inspiratory fraction of oxygen. Biochemistry values and arterial blood gases, blood count and coagulation parameters on admission to the ICU during the first 7 days from ICU admission. Pharmacological therapies received for COVID-19 disease during the ICU stay: azitromycin, corticosteroids, hydroxychloroquine, antiretrovirals (lopinavir/ritonavir), tocilizumab, oseltamivir, darunabir, remdesivir, baricitinib.

Bacterial / fungal infections acquired in the ICU (pneumonia, bacteriemia): isolated microorganisms in diagnostic samples, isolated microorganisms in surveillance samples (oropharynx and rectum if surveillance samples are available); antibiotic treatment.

Ventilatory management: prone positioning, administration of inhaled nitric oxide, performance of tracheostomy, date of tracheotomy, modality of tracheotomy (surgical, percutaneous).

Classification of predefined causes of death:

Refractory hypoxemia (peripheral oxygen saturation measured by pulse oximetry less than 80%, or PaO2 <60 mmHg of arterial blood sample) despite maximum ventilatory support (FiO2 100%, PEEP level> 5 cm H2O) with maintenance MAP> 60 mmHg in the 3 hours prior to exitus lethalis.

Refractory shock (mean arterial pressure less than 60 mmHg despite vasoactive support with norepinephrine at> 2 mcg / kg / min and / or dobutamine at> 20 microgr / kg / min, and serum lactate level> 2 mmol / L in the 3 hours prior to exitus lethalis), associated or not with organ failure, but with peripheral oxygen saturation measured by pulse oximetry greater than 90%, with no evidence of documented infection in the previous 48 hours.

Septic shock. A refractory shock which fulfill previous criteria plus the presence of a documented infection in the 48 hours prior to exitus lethalis.

Others: Pulmonary thromboembolism (defined based on clinical suspicion, associated with any of the classifications [Wells or Geneva] according to the low, intermediate or high probability and the determination of the high D-dimer (> 500 μg/L) in the 24 hours prior to exitus lethalis; Incohercible bleeding; Yatrogenic respiratory complications (accidental exit of the orotracheal tube with impossibility of obtaining an artificial airway, fatal obstruction of the orotracheal tube); Arrhythmias: sudden unanticipated onset of malignant arrhythmias (irreversible ventricular fibrillation), or asystole. Arrhythmias appearing during the last minutes before exitus lethalis will be excluded.

Main outcomes. ICU mortality, 28-day mortality, and hospital mortality. Secondary outcomes: appearance of nosocomial infections during ICU admission (ventilator-associated pneumonia , nosocomial pneumonia, catheter-related bacteremia, bacteraemia); development of complications during ICU admission (development of acute respiratory distress, barotrauma, development of organ failure [cardiovascular, renal, hepatic, hematological]), duration of mechanical ventilation, length of ICU stay, length of hospital stay, withdrawald of life support, and cause of mortality.

Statistic analysis. Given the estimated mortality of 40% of the cases hospitalized in the ICU, a convenience sample size of 600 participants will be estimated. Considering a loss of 15% for the outcomes, 750 subjects will finally be included.

To evaluate the risk factors associated with the mortality of critically ill patients with COVID-19, a logistic model adjusted for baseline variables (age, severity at ICU admission), empirical treatment received, failure of non-invasive respiratory support will be performed.

The effectiveness of empirical treatments for COVID-19 will be performed through logistic analysis adjusted for age, severity at admission and complications during ICU admission.

In addition, a stratified cluster analysis will be proposed for ICUs that apply the SDD strategy and units that do not routinely use SDD.

Data quality. The data will be reviewed and approved by the Steering Committee of the study and validated by the collaborating researcher responsible for each center. All data will be centrally reviewed. Alerts will be sent for lost data, aberrant data or discrepancies thereof.

At each center, local study investigators will review data from 5% of randomly selected participants, and all participants about whom evaluators may have questions about inconsistent data.

The data collection of all included cases will be verified by an independent research coordinator hired through an external CRO and who will evaluate the quality of data collection independently of the main researcher. Data collection will be re-evaluated until the forms and all results are completed.

Full data will be required to include subjects in the final analysis, and only subjects without missing data will be accepted for the primary variables or patients with missing data less than 10% for the secondary variables, if these cannot be retrieved by the investigators. All bizarre data will be sent to the reference centers for verification. The presence of missing data in the main variables will be reason for the exclusion of the participant in the analysis.

Ethical-legal aspects. The study will be carried out in accordance with the updated Helsinki declaration in its latest version. The study protocol, together with the data collection sheets and Annexes will be sent for approval to the Ethics and Research Committee of the University Hospital of Getafe, and will ask them for a waiver consent due to the characteristics of the study design (non-intervention study for statistical purposes, action plan to improve the quality of care, in a health emergency situation), as provided in the spanish laws.

This study does not include any control group. Participation in this study does not imply any risk for the included patients since it is based on the usual clinical practice in common use in all hospitals, which are already applied at the Getafe University Hospital.

The study will be based on the Spanish legislation for biomedical research, and in accordance with national laws of Protection of Personal Data and guarantee of them that the identity of the subject will be kept confidential and anonymous throughout the study, in such a way that no personal data will be collected that allows the identification of the subjects included and only the data necessary to achieve the study objectives will be collected.

Confidentiality The use, disclosure, publication or dissemination of the document is not authorized in any way without the written consent of the Steering Committee. Given that the study proposes the analysis of the usual clinical practice, it is considered not pertinent to contract a civil liability insurance, since it is a low-intensity clinical study.

During the period of inclusion of the participants, the database to which only the study coordinating team (principal investigator and co-investigators) will have access will be generated anonymously, with irreversible dissociation of personal data.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age who are admitted to the ICU with the confirmed diagnosis of COVID-19.

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case definition : Any critically ill patients with a positive respiratory tract sample result (tracheal aspirate or nasopharyngeal exudate) using the PCR9 technique for the SARS-CoV-2 virus and requiring admission to the ICU at trial will be considered a confirmed case of COVID-19 disease of the doctor responsible for the sick.
Sampling Method: Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
ICU mortality | events during the ICU stay, up to 3 months
  rate (%)

SECONDARY OUTCOMES:
hospital mortality | events through study completion during the hospital stay, up to 5 months
  rate (%)
28-day mortality | events through study completion considered from ICU admission up to 28 days
  rate (%)
effectiveness of treatment | through study completion considered from ICU admission until ICU discharge, up to 3 months
  rate (%). Incidence of outcome measures (ICU mortality), and appearance of complications (pneumonia or bacteriemia during ICU stay).
length of ICU stay | through study completion during ICU stay considered from ICU admission until ICU discharge as date of inclusion until the date of first documented discharge or date of death from any cause, whichever came first, assessed up to 3 months
  days
length of hospital stay | through study completion during ICU stay considered from ICU admission until ICU discharge as date of inclusion until the date of first documented hospital discharge or date of death from any cause, whichever came first, assessed up to 5 months
  days
ventilator-associated pneumonia | through duration of invasive ventilatory support period (from intubation date until date of successful extubation) through study completion up to 3 months
  rate (%)
bacteriemia | through study completion, up to 28-days
  rate (%)
barotrauma | through study completion, up to 28-days
  rate (%)
duration of mechanical ventilation | period of invasive controlled ventilatory support from date of orotraqueal intubation until date of successful extubation or assessed up to 3 months whichever came first
  days

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Peñuelas, P.h.D, Principal Investigator — Fundación de Investigación del Hospital Universitario de Getafe
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol, SAP
Time Frame: 3 months
Access Criteria: Direct request to the Principal Investigator

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Result] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Derived] Penuelas O, Del Campo-Albendea L, de Aledo ALG, Anon JM, Rodriguez-Solis C, Mancebo J, Vera P, Ballesteros D, Jimenez J, Maseda E, Figueira JC, Franco N, Algaba A, Aviles JP, Diaz R, Abad B, Canabal A, Abella A, Gordo F, Garcia J, Suarez JG, Cedeno J, Martinez-Palacios B, Manteiga E, Martinez O, Blancas R, Bardi T, Pestana D, Lorente JA, Muriel A, Esteban A, Frutos-Vivar F. Long-term survival of mechanically ventilated patients with severe COVID-19: an observational cohort study. Ann Intensive Care. 2021 Oct 2;11(1):143. doi: 10.1186/s13613-021-00929-y. PMID 34601646